CLINICAL TRIAL: NCT00375141
Title: Long-Pulsed Dye Laser and Intense Pulsed Light for Skin Rejuvenation.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion, treatments and follow-up are finished
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: KF-01-316279
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-06

CONDITIONS: Photodamaged Skin
MeSH Terms: interventions — Lasers, Dye

INTERVENTIONS:
Device: Pulsed dye laser, Intense pulsed light

SUMMARY:
The purpose of the trial is to compare clinical efficacy and occurrence of side effects in the treatment of photodamaged skin with Pulsed Dye Laser and Intense Pulsed Light.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate bilateral facial photodamage
* Symmetry in the facial area of wrinkles, skin texture, pigmentary changes and telangiectasia
* Fitzpatrick's skin type of Type I, II, or III, without significant tan
* Age > 40 years
* Able to read and comprehend Danish
* Informed consent agreement signed by the subject
* Willingness to follow the treatment schedule and posttreatment follow-up evaluations
* Willingness to allow photographs of the treated area to be taken for evaluation of efficacy.

Exclusion Criteria:

* Scarring or infection of the area to be treated
* Known photosensitivity
* Presence of a suntan in the area to be treated
* Subjects taken medication known to induce photosensitivity in the previous three months
* Known anticoagulation or thromboembolic conditions
* Subjects taking anticoagulation medication
* Subjects taking Accutane within the past 6 months
* Subjects treated with aspirins or anti-inflammatory drugs
* Subjects who are immunocompromised or have a medical history that is inappropriate for the study per the investigator's clinical judgment.
* Dermabrasion, chemical peel, laser or IPL treatment, or collagen injection therapy in the facial area in the past 12 months.
* Previous formation of hypertrophic scars or keloids
* Subjects who are pregnant or lactating
* Asymmetry in the facial area of wrinkles, skin texture, pigmentary changes and telangiectasia

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark